CLINICAL TRIAL: NCT00872742
Title: Acceptance Enhanced Behavior Therapy for Trichotillomania
Brief Title: Testing a New Therapy for Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Douglas Woods, Professor of Psychology, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH080966 (NIH); R01MH080966 (NIH); DATR A2-AIR; 1R01MH080966 (NIH); NIMH-3065236
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Trichotillomania
Keywords: Impulse Control Disorders; Behavior Therapy; Acceptance; Habit Reversal
MeSH Terms: conditions — Trichotillomania; Disruptive, Impulse Control, and Conduct Disorders | interventions — Acceptance and Commitment Therapy; Behavior Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive acceptance enhanced behavior therapy (AEBT) for trichotillomania (TTM).
  Interventions: Behavioral: Acceptance enhanced behavior therapy (AEBT)
- 2 (Active Comparator): Participants will receive psychoeducation and supportive therapy (PST) for TTM.
  Interventions: Behavioral: Psychoeducation and supportive therapy (PST)

INTERVENTIONS:
Behavioral: Acceptance enhanced behavior therapy (AEBT) — Ten 1-hour sessions over 12 weeks, enhancing awareness of hair-pulling behavior and teaching strategies to deal with hair pulling
  Other Names: Acceptance and Commitment Therapy; ACT; Habit Reversal; Behavior Therapy
  Arms: 1
Behavioral: Psychoeducation and supportive therapy (PST) — Ten 1-hour sessions over 12 weeks, teaching the participant about hair pulling and discussing how hair pulling affects those who do it
  Other Names: Supportive Therapy; Psychoeducation
  Arms: 2

SUMMARY:
This study will test the effectiveness of a new behavioral therapy for adults with trichotillomania (compulsive hair pulling).

DETAILED DESCRIPTION:
Trichotillomania (TTM) is a disorder in which people compulsively pull out their own hair. Treatments for TTM sometimes do not have long-term effectiveness. Acceptance and commitment therapy (ACT) is a therapeutic approach thought to have longer lasting effects than standard cognitive behavioral therapy (CBT) approaches, because ACT focuses on accepting thoughts and behaviors as opposed to changing them. Previous research indicates that a combination of ACT and habit reversal behavioral therapy is more effective than no treatment. This study will test whether a combination of ACT and behavioral therapy, called acceptance enhanced behavioral therapy (AEBT), is more effective than the current standard treatment for TTM.

Participation in this study will last 12 weeks, and follow-up assessments will last for 6 months. At study entry, participants will complete a brief intelligence test and an in-person interview about their medical history, psychiatric history, and hair pulling. At their second visit, participants will have digital pictures taken of their hair-pulling sites and complete two computer tasks measuring their response inhibition and cognitive flexibility. After the second visit, participants will be randomly assigned to receive either AEBT or psychoeducation and supportive therapy (PST)-a standard treatment for TTM. Both treatments will involve ten 1-hour sessions completed over 12 weeks. Assessments of participants will occur after 6 weeks of treatment, at treatment completion, and after 6 months. These assessments will measure treatment effectiveness, based on several clinical scales and measures of TTM symptoms. Participants who receive PST during this study will be offered AEBT afterward.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV diagnosis of trichotillomania
* Massachusetts General Hospital Hair Scale score greater than 12
* Wechsler Test of Adult Reading score greater than 85
* Fluent in English
* Outpatient status
* Agreement to not alter the dosage of any psychotropic medication throughout the course of the study, or, if such a dosage change is required, understanding that the participant will continue to receive treatment, and data will continue to be collected on him or her
* Individuals who eat their hair after pulling will be eligible for participation only after they have received a physical exam from their primary care physician to determine whether there is any gastrointestinal blockage due to hair pulling, which would require more immediate clinical care.

Exclusion Criteria:

* Diagnosis of bipolar disorder, psychotic disorder, mental retardation, pervasive developmental disorder, or current substance dependence (with the exception of nicotine dependence)
* Current mood or anxiety disorder with an active suicide risk
* Currently receiving psychotherapy for trichotillomania or another psychiatric condition
* Initiation or change in the dosage of any psychotropic medication for up to 8 weeks preceding participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions-Improvement Scale | Measured after 6 weeks, 12 weeks, and 6 months

SECONDARY OUTCOMES:
Massachusetts General Hospital Hairpulling Scale | Measured at screening, baseline, and after 6 weeks, 12 weeks, and 6 months
National Institute of Mental Health (NIMH) Trichotillomania Severity and Impairment Scales | Measured at screening, baseline, and after 6 weeks, 12 weeks, and 6 months
Clinical Global Impressions-Severity Scale | Measured at screening, baseline, and after 6 weeks, 12 weeks, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Woods, PhD, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Barber KE, Woods DW, Deckersbach T, Bauer CC, Compton SN, Twohig MP, Ricketts EJ, Robinson J, Saunders SM, Franklin ME. Neurocognitive functioning in adults with trichotillomania: Predictors of treatment response and symptom severity in a randomized control trial. Behav Res Ther. 2024 Aug;179:104556. doi: 10.1016/j.brat.2024.104556. Epub 2024 May 9. PMID 38761558
- [Derived] Houghton DC, McFarland CS, Franklin ME, Twohig MP, Compton SN, Neal-Barnett AM, Saunders SM, Woods DW. DSM-5 Trichotillomania: Perception of Adults With Trichotillomania After Psychosocial Treatment. Psychiatry. 2016 Summer;79(2):164-169. doi: 10.1080/00332747.2016.1144438. PMID 27724833